CLINICAL TRIAL: NCT06197438
Title: PD-1 Antibody(Tislelizumab) Plus Irinotecan Combined With POF in Treatment Naive Advanced Gastric Cancer: A Phase II Study.
Brief Title: Phase II Study of the Combination of Irinotecan and POF (POFI) and Tislelizumab in Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYLT-025
Record Dates: First submitted 2023-03-23; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — tislelizumab; Oxaliplatin; Levoleucovorin; Fluorouracil; Irinotecan; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- POFI and Tislelizumab (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Oxaliplatin; Drug: Levo-Leucovorin; Drug: 5-fluorouracil; Drug: Irinotecan Hydrochloride; Drug: Paclitaxel

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab will be administered on day 1 of each cycle at 200mg once every 21 days.
Drug: Oxaliplatin — Oxaliplatin will be administered on day 1 of each cycle at 85mg/m2 once every 14 days.
Drug: Levo-Leucovorin — Levo-Leucovorin will be administered on day 1 of each cycle at 200 mg/m2 once every 14 days.
Drug: 5-fluorouracil — 5-fluorouracil will be administered at 2400 mg/m2 over 46-hour every 14 days.
Drug: Irinotecan Hydrochloride — Irinotecan will be administered on day 1 of each cycle at 135 mg/m2 once every 14 days.
Drug: Paclitaxel — Paclitaxel will be administered on day 1 of each cycle at 90 mg/m2 once every 14 days.

SUMMARY:
This study is a single center, phase II study, to evaluate the effectiveness and safety of PD-1 Antibody(Tislelizumab) Plus Irinotecan Combined With POF(paclitaxel plus oxaliplatin plus 5-fluorouracil plus leucovorin) , in the first-line treatment for patients with advanced/metastatic gastric cancer.

DETAILED DESCRIPTION:
This is a exploratory, single-arm, open-label trial. The investigator's primary purpose is to compare that ORR of patients with Tislelizumab plus Irinotecan and POF for advanced/metastatic gastric cancer.

In treatment period, patients will be administrated Tislelizumab plus Irinotecan and POF, every 21 days for 1 cycle, until disease progression, toxicity intolerance, withdrawal of informed consent, patients judged must be terminated study termination.

The imaging evaluation was performed according to the RECIST 1.1 criteria every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced unresectable, histologically confirmed adenocarcinoma of the gastric or gastroesophageal junction.
2. With or without measurable lesions.
3. Patients must have a performance status of 0-1 on the Eastern Cooperative Oncology Group (ECOG) scale.
4. Without serious system dysfunction and could tolerate chemotherapy. With normal marrow, liver and renal function: a hemoglobin (HGB) of ≥100g/L (without blood transfusion during 14 days); a leucopenia count of ≥4.0×109/L; a platelet count of ≥100×109/L; a total bilirubin (TBil) of ≤1.5 upper normal limitation (UNL); a creatinine (Cr) of ≤ 1.5 UNL; a creatinine clearance rate ≥ 50ml/min (Cockcroft-Gault); a alanine aminotransferase (ALAT) and aspartate aminotransferase (ASAT) of ≤2.5 UNL or ≤5 UNL in case of liver metastasis.
5. Life expectancy ≥3 months.
6. With normal electrocardiogram results and no history of congestive heart failure.
7. With normal coagulation function: activated partial thromboplastin time (APTT), prothrombin time (PT) and INR, each ≤ 1.5 x ULN.
8. Female subjects of child-bearing potential must agree to use contraceptive measures starting 1 week before the administration of the first dose of Tislelizumab until 8 weeks after discontinuing study drug. Male subjects must agree to use contraceptive measures during the study and 8 weeks after last dose of study drug
9. With written informed consent signed voluntarily by patients themselves or their supervisors witted by doctors.
10. With good compliance and agree to accept follow-up of disease progression and adverse events.

Exclusion Criteria:

1. Patients with a history of another neoplastic disease within the past three years, excluding basal cell carcinoma of the skin, cervical carcinoma in situ, or nonmetastatic prostate cancer.
2. Patients with brain or central nervous system metastases, including leptomeningeal disease.
3. Pregnant (positive pregnancy test) or breast feeding.
4. Serious, non-healing wound, ulcer, or bone fracture.
5. Significant cardiac disease as defined as: unstable angina, New York Heart 6.Association (NYHA) grade II or greater, congestive heart failure, history of myocardial infarction within 6 months Evidence of bleeding diathesis or coagulopathy.

7.History of a stroke or CVA within 6 months. 8.Clinically significant peripheral vascular disease. 9.Inability to comply with study and/or follow-up procedures. Patients with any other medical condition or reason, in that investigator's opinion, makes the patient unstable to participate in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-04-11 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | From enrollment to 12 month
  ORR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR. ORR was assessed by the investigator according to RECIST version 1.1 and is based on BOR, which is defined as best response recorded from start of study treatment until disease progression/recurrence or death. Participants needed to have two consecutive assessments of PR or CR to be a responder. Only participants with measurable disease at baseline were included in the analysis of BOR and who did not have any evaluable post-baseline assessments were classified as not evaluable.The ORR will be reported by percentage with each arms and appropriate confidence intervals.

SECONDARY OUTCOMES:
1.Progression-Free Survival(PFS) | From enrollment to 12 month
  PFS was defined as the time from randomization to first documented disease progression (PD) using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) or death from any cause, whichever occurred first. For target lesions, PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions.The PFS will be will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median PFS, hazard ratio with appropriate confidence intervals will be reported.The PFS will be will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median PFS, hazard ratio with appropriate confidence intervals will be reported.
Overall Survival (OS) | From enrollment to 12 month
  Overall Survival (OS), defined as the time from the date of randomization to the date of death, regardless of the cause of death. Participants who were alive at the time of the analysis were censored at the date of the last follow-up assessment. Participants without follow-up assessment were censored at the day of last study medication and participants with no post-baseline information were censored at the date of randomization.The OS will be will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median OS, hazard ratio with appropriate confidence intervals will be reported.
Disease control rate(DCR) | From enrollment to 12 month
  DCR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR or SD. ORR was assessed by the investigator according to RECIST version 1.1 and is based on BOR, which is defined as best response recorded from start of study treatment until disease progression/recurrence or death. Participants needed to have two consecutive assessments of PR or CR or SD to be a responder. Only participants with measurable disease at baseline were included in the analysis of BOR and who did not have any evaluable post-baseline assessments were classified as not evaluable.The ORR will be reported by percentage with each arms and appropriate confidence intervals.

IPD SHARING:
Plan to Share IPD: No